CLINICAL TRIAL: NCT00746421
Title: Phase IV Study of Quetiapine XR Aimed at Disability and Cognitive Impairments.
Brief Title: Quetiapine XR for Cognitive and Functional Disability in Clinically Stable Patients With Bipolar Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdrew funding
Sponsor: Emory University (Other)
Collaborators: Duke University (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Jeffrey Rakofsky, Assistant Professor of Psychiatry and Behavioral Sciences, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00009874
Record Dates: First submitted 2008-09-03; First posted 2008-09-04 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar Disorder; Cognitive Impairment
Keywords: Cognition; attention; bipolar; disability
MeSH Terms: conditions — Bipolar Disorder; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Quetiapine XR 200-400 mg/day
  Interventions: Drug: Quetiapine XR
- 2 (Placebo Comparator): Placebo one pill per day matching 200, 300, or 400 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine XR — oral doses, 200 mg, 300 mg, 400 mg
  Other Names: Seroquel XR
  Arms: 1
Drug: Placebo — 200mg, 300mg or 400mg
  Arms: 2

SUMMARY:
Quetiapine has been reported to have beneficial cognitive effects in several randomized controlled trials in schizophrenia. It has not yet been studied in bipolar disorder, but promising results from the use of extended release quetiapine for the maintenance treatment of bipolar disorder suggests that its cognitive benefits could be detected. Moreover, quetiapine has been shown to have direct beneficial effects on performance-based measures of social competence in schizophrenia and to improve quality of life (QoL) in bipolar depression. The investigators propose to study quetiapine augmentation of mood stabilizer monotherapy in clinically stable patients with bipolar disorder. This will be a randomized, placebo controlled trial, with attentional impairments as the primary outcome and other cognitive performance variables and measures of social and everyday living skills, as well as subjective QoL, as the secondary outcomes.

DETAILED DESCRIPTION:
In contrast to previous conceptions of bipolar disorder as an illness where cognitive impairments were limited to manic and depressed episodes, it has become clear that cognitive impairments are common in clinically stable bipolar patients.

Quetiapine has been reported to have beneficial cognitive effects in several randomized controlled trials in schizophrenia. It has not yet been studied in bipolar disorder, but promising results from the use of extended release quetiapine for the maintenance treatment of bipolar disorder suggests that its cognitive benefits could be detected. Moreover, quetiapine has been shown to have direct beneficial effects on performance-based measures of social competence in schizophrenia and to improve quality of life (QoL) in bipolar depression. We propose to study quetiapine augmentation of mood stabilizer monotherapy in clinically stable patients with bipolar disorder. This will be a randomized, placebo controlled trial, with attentional impairments as the primary outcome and other cognitive performance variables and measures of social and everyday living skills, as well as subjective QoL, as the secondary outcomes.

An additional possible benefit of quetiapine treatment, and one that is directly relevant to neuropsychological performance, is that of increased activity of cortical norepinephrine (NE). Thus, in studies of cognitive enhancement with quetiapine, examination of cortical NE neet occupancy will be of substantial interest.

General Background: This will be a three site study which will include Emory University (Coordinating site), Duke University, and University of Toronto. We choose to have three sites so that the difficult task of recruiting clinically stable patients with bipolar can be accomplished quickly and the study can be completed within a two-year time frame.

Subjects: We will recruit 100 patients for this study. Fifty percent of them will receive active treatment with quetiapine XR. All participants will meet diagnostic criteria for bipolar I and II disorder and have medical record-based evidence of at least one previous manic or mixed episode. They will be clinically stable, as evidence by meeting criteria for low scores on both the Young Mania Rating Scale (YMRS) and the Montgomery-Asberg Depression rating scale (MADRS). They will also be receiving therapy with mood stabilizers, either lithium or an approved mood stabilizing agent.

Visit Schedule: This is a 10 week study with a six-week active treatment protocol. All interested patients who meet study entry criteria will be screened for stability four and two weeks prior to the baseline assessment. Patients will also be re-assessed for stability at baseline. Patients who fail to meet entry criteria at baseline can come back for a second screening after 2 and 4 weeks.

Throughout treatment, medication adjustments will be limited to changes of less than 25% during this time period.

Assessments: Cognitive assessments will be performed at baseline, week 2 and week 6 of active treatment.

Clinical Assessments will be performed at screening and rescreening, baseline, weeks 2 and 6.

Biological Measures: Bloods for NE net occupancy will be drawn at baseline, week 2, and week 6. Serum levels of quetiapine at all three assessments will also be examined.

Cognitive Assessments:

We will focus our cognitive assessment on the types of cognitive impairments previously reported in bipolar disorder. Our focus will be on attention, episodic memory, processing speed, and working memory. This same instrumentation has proven able to detect sedation as well, so that we can use the results of our assessment to identify any potential adverse sedation effects.

ELIGIBILITY:
Inclusion criteria:

1. Provision of written informed consent
2. A primary diagnosis of Bipolar disorder type 1 or 2, with a definite history of manic or hypomanic episodes by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV).
3. Females and/or males aged 18-65 years.
4. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment.
5. Able to understand and comply with the requirements of the study.
6. YMDRS score <13.
7. MADRS score <19.
8. Currently receiving medication therapy with lithium, valproate, or lamotrigine or any combination thereof. (preference given to lithium and/or valproate).
9. Clinically stable for 4 weeks prior to study entry, confirmed at week 2.

Exclusion criteria:

1. Intolerance of quetiapine
2. Change in mood stabilizer medication or dose in the last 4 weeks, change in antidepressant medication or dose in the last two months.
3. Current treatment with carbamazepine, stimulants, atomoxetine, or another antipsychotic
4. Current treatment with norepinephrine reuptake inhibiting antidepressants (Milnacipran, bupropion, paroxetine, duloxetine, venlafaxine, all MAOI's, all TCAs)
5. Current pregnancy or lactation
6. Active Anorexia nervosa or Bulimia nervosa in the past six months
7. History of non-affective psychotic disorders (including schizoaffective disorder)
8. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
9. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
10. Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
11. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
12. Active Substance/ alcohol abuse or dependence in the past three months before enrollment ( except for caffeine or nicotine dependence), as defined by DSM-IV criteria Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
13. Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hyperlipidemia, hypertension) as judged by the investigator
14. Involvement in the planning and conduct of the study
15. Previous enrolment or randomisation of treatment in the present study.
16. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
17. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrollment glycosylated hemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomization. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
18. An absolute neutrophil count (ANC) of < 1.5 x 10^9 per liter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Rakofsky, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - Duke University, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period continued until April 2012 and occurred in medical clinics and through advertisements.
Pre-assignment Details: There was a run-in period to ensure mood stability before randomization. Some patients were lost to follow up during this period.
Groups:
- Quetiapine XR Group: Quetiapine XR 200-400 mg/day
- Placebo Group: Placebo one pill per day matching 200, 300, or 400 mg active medications
Period: Overall Study
Arm/Group | Quetiapine XR Group | Placebo Group
Started | 12 | 11
Completed | 5 | 9
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR Group | Placebo Group | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (14.9) | 42.6 (13.9) | 40 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Continuous Performance Test-Identical Pairs Version
Description: The Continuous Performance Test, Identical Pairs version (CPT-IP) is a cognitive test that requires a subject to respond whenever two identical stimuli appear in a row within a sequence of 150 rapidly flashed trials. The outcome is measured as d' (detection signal) and is dimensionless. Among healthy adult men and women, d' scores ranged from 3.07-4.57 (Chen et al. Schizophrenia Bulletin, 1998; 24(1):163-174). The higher the value the better the performance. The d' is calculated by averaging the d' scores from three trials.
Time Frame: 6 weeks
Population: The statistical analysis was planned as Intention to treat with LOCF as the endpoint variable. We initially aimed to enroll 50 patients per group but because the study was terminated early, with a total of only 32 subjects. These numbers are too small to have a meaningful statistical outcome and so this between group comparison was not performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Quetiapine XR Group | Placebo Group
Number analyzed (Participants) | 5 | 9
units on a scale | 2.5 (0.82) | 2.8 (0.83)

2. Secondary Outcome: Brief Assessment of Cognition for Affective Disorders (BAC-A)
Description: This is a series of neurocognitive tests and includes brief assessments of attention, motor speed, working memory, verbal memory, reasoning and problem solving, verbal fluency, affective interference, and emotion inhibition. The total BAC-A score is represented by a composite T-score which is dimensionless. This is computed by adding up the scores for each trial of a test domain (e.g. verbal memory) within the cognitive battery. Each test domain total is then inputted into a proprietary BAC-A calculator which determines the composite T-scores. A higher score indicates better performance. A study of 404 healthy adults demonstrated a mean composite score of 50 with a standard deviation of 10 (Keefe et al. Schizophrenia Bulletin. 2008; 102: 108-115).
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale (composite t-score)
Arm/Group | Quetiapine XR Group | Placebo Group
Number analyzed (Participants) | 5 | 9
units on a scale (composite t-score) | 49.6 (12.1) | 47.8 (11.5)

ADVERSE EVENTS:
Arm/Group | Quetiapine XR Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 10/12 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine XR Group (N=12) | Placebo Group (N=11)
sedation (Psychiatric disorders) | 10 (10) | 0 (0)

LIMITATIONS AND CAVEATS:
We were unable to perform the pre-planned primary and secondary statistical analyses between group comparisons as the groups sizes were too small to compare meaningfully.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less